CLINICAL TRIAL: NCT03997383
Title: APOLLO-B: A Phase 3, Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Efficacy and Safety of Patisiran in Patients With Transthyretin Amyloidosis With Cardiomyopathy (ATTR Amyloidosis With Cardiomyopathy)
Brief Title: APOLLO-B: A Study to Evaluate Patisiran in Participants With Transthyretin Amyloidosis With Cardiomyopathy (ATTR Amyloidosis With Cardiomyopathy)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-TTR02-011; 2019-001458-24 (EudraCT Number)
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin Amyloidosis (ATTR) With Cardiomyopathy
Keywords: RNAi therapeutic; Transthyretin; TTR; Amyloidosis; Cardiomyopathy; ATTR
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis; Cardiomyopathies | interventions — patisiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patisiran (Experimental): Participants will be administered multiple doses of patisiran in the double-blind and open-label extension period.
  Interventions: Drug: Patisiran
- Placebo (Placebo Comparator): Participants will be administered multiple doses of placebo in the double-blind period. In the open-label extension period, participants will be administered multiple doses of patisiran.
  Interventions: Drug: Placebo; Drug: Patisiran

INTERVENTIONS:
Drug: Placebo — Normal saline (0.9% NaCl) matching volume of patisiran doses will be administered intravenously.
  Arms: Placebo
Drug: Patisiran — Patisiran will be administered by intravenous (IV) infusion.
  Other Names: ALN-TTR02; patisiran-lipid nanoparticle (LNP)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of patisiran in participants with ATTR amyloidosis with cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of ATTR amyloidosis with cardiomyopathy, classified as either hereditary ATTR amyloidosis with cardiomyopathy or wild-type ATTR amyloidosis with cardiomyopathy
* Medical history of heart failure with at least 1 prior hospitalization for heart failure, or current clinical evidence (signs and symptoms of heart failure)
* Clinically stable with no cardiovascular related hospitalizations within 6 weeks of study start
* Has never taken tafamidis before (tafamidis naïve) or currently on tafamidis for ≥6 months with evidence of disease progression while on tafamidis treatment
* Able to complete ≥150 m on the 6-minute walk test
* Screening N-terminal pro B-type natriuretic peptide (NT-proBNP), a blood marker of heart failure severity, >300 ng/L and <8500 ng/L; in participants with permanent or persistent atrial fibrillation, screening NT-proBNP> 600 ng/L and <8500 ng/L

Exclusion Criteria:

* Known primary amyloidosis (AL) or leptomeningeal amyloidosis.
* Received prior TTR lowering treatment
* New York Heart Association heart failure classification of III and at high risk
* New York Heart Association heart failure classification of IV
* Neuropathy requiring cane or stick to walk, or is wheelchair bound
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2
* Abnormal liver function
* Has hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Has non-amyloid disease that significantly affects ability to walk (e.g., severe chronic obstructive pulmonary disease, severe arthritis, or peripheral vascular disease affecting ambulation)
* Prior or planned heart, liver, or other organ transplant
* Other cardiomyopathy not related to ATTR amyloidosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2027-03-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (83):
- United States (17):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Skokie, Illinois
  - Clinical Trial Site, Iowa City, Iowa
  - Clinical Trial Site, Kansas City, Kansas
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Burlington, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Norfolk, Virginia
- Argentina (6):
  - Clinical Trial Site, Buenos Aires, Buenos Aires
  - Clinical Trial Site, San Juan Bautista, Buenos Aires
  - Clinical Trial Site, Córdoba, Córdoba Province
  - Clinical Trial Site, Rosario, Santa Fe Province
  - Clinical Trial Site, Santa Fe, Santa Fe Province
  - Clinical Trial Site, Buenos Aires
- Australia (3):
  - Clinical Trial Site, Westmead, New South Wales
  - Clinical Trial Site, Woolloongabba, Queensland
  - Clinical Trial Site, Box Hill, Victoria
- Belgium (4):
  - Clinical Trial Site, Liège, LIE
  - Clinical Trial Site, Hasselt, LIM
  - Clinical Trial Site, Aalst, OVL
  - Clinical Trial Site, Roeselare, WVL
- Brazil (5):
  - Clinical Trial Site, Porto Alegre, Rio Grande do Sul
  - Clinical Trial Site, Ribeirão Preto, São Paulo
  - Clinical Trial Site, São Paulo, São Paulo
  - Clinical Trial Site, Rio de Janeiro
  - Clinical Trial Site, São Paulo
- Bulgaria (3):
  - Clinical Trial Site, Sofia, Sofia-Grad
  - Clinical Trial Site, Sofia
  - Clinical Trial Site, Stara Zagora
- Clinical Trial Site, Santiago, Chile
- Czechia (3):
  - Clinical Trial Site, Prague, Praha, Hlavní Mesto
  - Clinical Trial Site, Brno
  - Clinical Trial Site, Prague
- Denmark (3):
  - Clinical Trial Site, Aarhus N, Aarhus
  - Clinical Trial Site, Copenhagen
  - Clinical Trial Site, Odense C
- France (4):
  - Clinical Trial Site, Clichy, Paris
  - Clinical Trial Site, Créteil, Val-de-Marne
  - Clinical Trial Site, Rennes
  - Clinical Trial Site, Toulouse
- Clinical Trial Site, Lai Chi Kok, Hong Kong
- Italy (4):
  - Clinical Trial Site, Bologna, Emilia-Romagna
  - Clinical Trial Site, Messina, Sicily
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Pavia
- Japan (7):
  - Clinical Trial Site, Nagoya, Aichi-ken
  - Clinical Trial Site, Kurume, Fukuoka
  - Clinical Trial Site, Matsumoto, Nagano
  - Clinical Trial Site, Suita, Osaka
  - Clinical Trial Site, Bunkyo-ku, Tokyo
  - Clinical Trial Site, Fukuoka
  - Clinical Trial Site, Kumamoto
- Clinical Trial Site, Mexico City, Mexico
- Netherlands (2):
  - Clinical Trial Site, Groningen
  - Clinical Trial Site, Maastricht
- New Zealand (2):
  - Clinical Trial Site, Christchurch
  - Clinical Trial Site, Hamilton
- Poland (4):
  - Clinical Trial Site, Lódz, Lódzkie
  - Clinical Trial Site, Warsaw, Masovian Voivodeship
  - Clinical Trial Site, Gdansk, Pomeranian Voivodeship
  - Clinical Trial Site, Katowice, Silesian Voivodeship
- Portugal (3):
  - Clinical Trial Site, Porto
  - Clinical Trial Site, Senhora da Hora
  - Clinical Trial Site, Viseu
- Clinical Trial Site, Seoul, South Korea
- Clinical Trial Site, Stockholm, Sweden
- Clinical Trial Site, Taipei, Taiwan
- United Kingdom (7):
  - Clinical Trial Site, Bellshill, Lanarkshire
  - Clinical Trial Site, London, London, City of
  - Clinical Trial Site, Hexham, Northumberland
  - Clinical Trial Site, Birmingham, West Midlands
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.

REFERENCES:
- [Derived] Mesquita CT, Schwartzmann P, Correia EB, Simoes MV, Biolo A, Duque DR, Jay PY, Fernandes F. Patisiran Treatment in the Brazilian Subpopulation of the Phase 3 APOLLO-B Study in Transthyretin Amyloidosis with Cardiomyopathy: Post Hoc Analysis. Arq Bras Cardiol. 2025 Mar;122(4):e20240568. doi: 10.36660/abc.20240568. English, Portuguese. PMID 40243852
- [Derived] Maurer MS, Kale P, Fontana M, Berk JL, Grogan M, Gustafsson F, Hung RR, Gottlieb RL, Damy T, Gonzalez-Duarte A, Sarswat N, Sekijima Y, Tahara N, Taylor MS, Kubanek M, Donal E, Palecek T, Tsujita K, Tang WHW, Yu WC, Obici L, Simoes M, Fernandes F, Poulsen SH, Diemberger I, Perfetto F, Solomon SD, Di Carli M, Badri P, White MT, Chen J, Yureneva E, Sweetser MT, Jay PY, Garg PP, Vest J, Gillmore JD; APOLLO-B Trial Investigators. Patisiran Treatment in Patients with Transthyretin Cardiac Amyloidosis. N Engl J Med. 2023 Oct 26;389(17):1553-1565. doi: 10.1056/NEJMoa2300757. PMID 37888916

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (DB)/Patisiran (OLE): Participants were administered placebo IV every 3 weeks during the 12-month double-blind (DB) treatment period. Participants will be administered patisiran 0.3 mg/kg IV every 3 weeks during the 36-month open label extension (OLE) period.
- Patisiran (DB+OLE): Participants were administered patisiran 0.3 mg/kg intravenously (IV) every 3 weeks during the 12-month DB treatment period. Participants will be administered patisiran 0.3 mg/kg IV every 3 weeks during the 36-month OLE period.
Period: Double-blind Treatment Period
Arm/Group | Placebo (DB)/Patisiran (OLE) | Patisiran (DB+OLE)
Started | 179 | 181
Treated | 178 | 181
Completed | 166 | 168
Not Completed | 13 | 13
Not completed — Adverse Event | 4 | 3
Not completed — Death | 4 | 4
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 3 | 6
Period: Open-label Extension Period
Arm/Group | Placebo (DB)/Patisiran (OLE) | Patisiran (DB+OLE)
Started | 166 | 168
Completed | 0 | 0
Not Completed | 166 | 168
Not completed — Ongoing | 148 | 151
Not completed — Adverse Event | 4 | 1
Not completed — Death | 8 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Subject Stopped Participation in the Study | 3 | 6
Not completed — Reason Not Specified | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS): All randomized participants who received any amount of study drug. Participants were summarized according to the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (DB)/Patisiran (OLE) | Patisiran (DB+OLE) | Total
Number analyzed (Participants) | 178 | 181 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (7.8) | 75.3 (6.5) | 74.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 160 | 161 | 321
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 15 | 23 | 38
  Black or African American | 15 | 16 | 31
  White | 140 | 138 | 278
  Other | 4 | 3 | 7
  Not Reported | 4 | 1 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 20 | 21 | 41
  Not Hispanic or Latino | 150 | 153 | 303
  Not Reported | 4 | 5 | 9
  Unknown | 4 | 2 | 6
6 Minute Walk Test (6MWT) [Median (Full Range); unit: meters] | 367.7 [130.0 to 740.0] | 356.8 [155.7 to 755.7] | 362.0 [130.0 to 755.7]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Month 12 in Six-Minute Walk Test (6-MWT)
Description: Distance in meters walked in 6 minutes, longer distances indicate greater functional capacity. Missing 6MWT values due to non-COVID-19 death or inability to walk due to ATTR disease progression were imputed using the worst 10th percentile change observed in the DB period. Missing 6-MWT values due to other reasons are multiply imputed to create 100 complete datasets. The change from baseline is averaged across the 100 complete datasets.
Time Frame: Baseline, Month 12
Population: Full Analysis Set: All randomized participants who received any amount of study drug. Participants were analyzed according to the treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: meters
Arm/Group | Placebo (DB)/Patisiran (OLE) | Patisiran (DB+OLE)
Number analyzed (Participants) | 178 | 181
meters | -21.345 [-68.268 to 12.750] | -8.150 [-54.651 to 29.510]
Statistical Analysis 1: Comparison: Placebo (DB)/Patisiran (OLE) vs Patisiran (DB+OLE); Test type: Superiority; p = 0.0162, Wilcoxon Rank Sum Test — P-value was determined by the Wilcoxon Rank Sum test,stratified by baseline tafamidis use.Analysis was performed on the 100 multiply-imputed datasets; Median Difference (Net) = 14.693, 95% CI 2-sided [0.693 to 28.692] — Median difference estimated by the Hodges-Lehmann method, stratified by baseline tafamidis use. Analysis was performed on the 100 multiply-imputed datasets

2. Secondary Outcome: Change From Baseline at Month 12 in Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ-OS) Score
Description: The KCCQ is a 23-item self-administered questionnaire quantifying 6 domains (symptoms, physical function, quality of life, social limitation, self-efficacy, and symptom stability) and 2 summary scores (clinical and overall summary [OS]). Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline, Month 12
Population: Full Analysis Set: All randomized participants who received any amount of study drug. Participants were analyzed according to the treatment to which they were randomized. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis at the specified timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (DB)/Patisiran (OLE) | Patisiran (DB+OLE)
Number analyzed (Participants) | 164 | 170
score on a scale | -3.396 (1.356) | 0.478 (1.363)
Statistical Analysis 1: Comparison: Placebo (DB)/Patisiran (OLE) vs Patisiran (DB+OLE); Test type: Superiority; p = 0.0397, MMRM — P-value was analyzed using mixed model repeated measures (MMRM) as described in the Statistical analysis plan; Least squares (LS) mean difference = 3.709, 95% CI 2-sided [0.176 to 7.242], Standard Error of Mean 1.796

3. Secondary Outcome: Composite Endpoint of All-Cause Mortality, Frequency of Cardiovascular (CV) Events (CV Hospitalizations and Urgent Heart Failure [HF] Visits) and Change From Baseline in 6-MWT Analyzed by Win Ratio
Description: The composite endpoint was analyzed using the stratified win ratio method, stratified by baseline tafamidis use. This method combines all-cause mortality, frequency of CV events (CV hospitalizations and HF visits) and change from baseline in 6-MWT in a hierarchical fashion. This method makes within-stratum pairwise comparisons for all patisiran-placebo participant pairs in a sequential manner (first mortality, then CV events, then 6-MWT), with later steps evaluated only in the case of a tie on the prior step. Within each stratum, the win ratio is the total number of 'winners' divided by the total number of 'losers' in the active group. A win ratio >1 represents a favorable outcome for patisiran.
Time Frame: Up to Month 12
Population: Participants from the Full Analysis Set (all randomized participants who received any amount of study drug (either placebo or patisiran), grouped based on their use of tafamidis at Baseline as pre-specified in the study protocol.
Measure: Number (95% Confidence Interval); unit: win ratio
Groups:
- Baseline Tafamidis: Participants from either the placebo or patisiran groups in DB period who were receiving treatment with tafamidis at Baseline.
- No Baseline Tafamidis: Participants from either the placebo or patisiran groups in DB period who were not receiving treatment with tafamidis at Baseline.
Arm/Group | Baseline Tafamidis | No Baseline Tafamidis
Number analyzed (Participants) | 91 | 268
win ratio | 1.22 [0.76 to 1.95] | 1.28 [0.97 to 1.70]
Statistical Analysis 1: Comparison: Baseline Tafamidis vs No Baseline Tafamidis; Test type: Superiority; p = 0.0574, Z-test; P-value was analyzed by a z-test using the mean and variance of the log-transformed win ratio estimate; Stratified Win Ratio = 1.27, 95% CI 2-sided [0.99 to 1.61]

4. Secondary Outcome: Composite Endpoint of All-Cause Mortality and Frequency of All-Cause Hospitalizations and Urgent HF Visits in Participants Not on Tafamidis at Baseline
Description: The hazard rate of all-cause mortality and all-cause hospitalizations and urgent HF visits will be compared between treatment groups using an Andersen-Gill model. A hazard ratio <1 represents a favorable outcome for patisiran.
Time Frame: Up to Month 12
Population: Participants from the Full Analysis Set [all randomized participants who received any amount of study drug (placebo or patisiran)] and were not receiving tafamidis at Baseline were included in the data analysis for the outcome measure as pre-specified in the study protocol.
Measure: Number; unit: hazard ratio
Groups:
- No Baseline Tafamidis: Participants from the placebo and the patisiran group in DB period who were not receiving treatment with tafamidis at Baseline.
Arm/Group | No Baseline Tafamidis
Number analyzed (Participants) | 268
hazard ratio | 0.997
Statistical Analysis 1: Comparison: No Baseline Tafamidis; Test type: Superiority; p = 0.9888, Andersen-Gill; Hazard Ratio (HR) = 0.997, 95% CI 2-sided [0.620 to 1.602] — HR was derived using an Andersen-Gill model, including the treatment arm, type of ATTR amyloidosis, baseline New York Heart Association (NYHA) class, and age as covariates

5. Secondary Outcome: Composite Endpoint of All-cause Mortality and Frequency of All-cause Hospitalizations and Urgent HF Visits in All Participants
Description: The hazard rate of all-cause mortality and all-cause hospitalizations and urgent HF visits was compared between treatment groups using a modified Andersen-Gill model. A hazard ratio <1 represents a favorable outcome for patisiran.
Time Frame: Up to Month 12
Population: All the participants from the Full Analysis Set [all randomized participants who received any amount of study drug (either placebo or patisiran)] were included in the data analysis for the outcome measure as pre-specified in the study protocol.
Measure: Number; unit: hazard ratio
Groups:
- All Participants: Participants were administered placebo or patisiran IV every 3 weeks during the 12-month double-blind (DB) treatment period. Participants will be administered patisiran 0.3 mg/kg IV every 3 weeks during the 36-month open label extension (OLE) period.
Arm/Group | All Participants
Number analyzed (Participants) | 359
hazard ratio | 0.883
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.5609, Modified Andersen-Gill; P-value was derived using the modified Andersen-Gill model stratified by baseline tafamidis use; Hazard Ratio (HR) = 0.883, 95% CI 2-sided [0.582 to 1.341] — HR was derived using the modified Andersen-Gill model stratified by baseline tafamidis use, including treatment arm, type of ATTR amyloidosis, baseline NYHA class, and age as covariates

ADVERSE EVENTS:
Time Frame: All-cause mortality: From the first dose of study drug up to data cut-off (approximately 17.5 months); Adverse events: From the first dose of study drug up to the end of double-blind treatment period (approximately 12 months)
Description: Deaths and adverse events collected during the double-blind treatment period were reported. Open-label extension (OLE) period of the study is ongoing and the results will be posted after study completion. In all-cause mortality, all deaths occurred in study due to any cause are reported.
Groups:
- Double-blind Period: Placebo: Participants were administered placebo IV every 3 weeks during the 12-month double-blind (DB) treatment period.
- Double-blind Period: Patisiran: Participants were administered patisiran 0.3 mg/kg intravenously (IV) every 3 weeks during the 12-month DB treatment period.
- Open Label Extension Period: Placebo (in DB Period) to Patisiran: Participants who received placebo in DB period will be administered patisiran 0.3 mg/kg IV every 3 weeks during the 36-month open label extension (OLE) period.
- Open Label Extension Period: Patisiran (in DB Period) to Patisiran: Participants who received patisiran in DB period will be administered patisiran 0.3 mg/kg IV every 3 weeks during the 36-month OLE period.
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Patisiran | Open Label Extension Period: Placebo (in DB Period) to Patisiran | Open Label Extension Period: Patisiran (in DB Period) to Patisiran
All-Cause Mortality (participants affected / at risk) | 8/178 | 4/181 | 10/166 | 9/168
Serious Adverse Events (participants affected / at risk) | 63/178 | 61/181 | 0/166 | 0/168
Other Adverse Events (participants affected / at risk) | 168/178 | 165/181 | 0/166 | 0/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Period: Placebo (N=178) | Double-blind Period: Patisiran (N=181) | Open Label Extension Period: Placebo (in DB Period) to Patisiran (N=166) | Open Label Extension Period: Patisiran (in DB Period) to Patisiran (N=168)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | NA | NA
Angina unstable (Cardiac disorders) | 1 | 0 | NA | NA
Atrial fibrillation (Cardiac disorders) | 4 | 5 | NA | NA
Atrial flutter (Cardiac disorders) | 0 | 2 | NA | NA
Atrioventricular block (Cardiac disorders) | 0 | 1 | NA | NA
Atrioventricular block complete (Cardiac disorders) | 4 | 2 | NA | NA
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | NA | NA
Atrioventricular block second degree (Cardiac disorders) | 2 | 0 | NA | NA
Bradycardia (Cardiac disorders) | 0 | 2 | NA | NA
Cardiac amyloidosis (Cardiac disorders) | 0 | 1 | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 1 | NA | NA
Cardiac failure (Cardiac disorders) | 13 | 15 | NA | NA
Cardiac failure acute (Cardiac disorders) | 2 | 1 | NA | NA
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | NA | NA
Chronotropic incompetence (Cardiac disorders) | 0 | 1 | NA | NA
Conduction disorder (Cardiac disorders) | 1 | 0 | NA | NA
Coronary artery disease (Cardiac disorders) | 3 | 0 | NA | NA
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 1 | NA | NA
Pericarditis (Cardiac disorders) | 1 | 0 | NA | NA
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | NA | NA
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | NA | NA
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | NA | NA
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | NA | NA
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | NA | NA
Enteritis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | NA | NA
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | NA | NA
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | NA | NA
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | NA | NA
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Asthenia (General disorders) | 1 | 0 | NA | NA
Chest discomfort (General disorders) | 1 | 0 | NA | NA
Chest pain (General disorders) | 3 | 0 | NA | NA
Infusion site phlebitis (General disorders) | 0 | 1 | NA | NA
Pyrexia (General disorders) | 1 | 0 | NA | NA
Vessel puncture site haematoma (General disorders) | 1 | 0 | NA | NA
Cholangitis (Hepatobiliary disorders) | 1 | 0 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | NA | NA
Amyloidosis (Immune system disorders) | 4 | 1 | NA | NA
Drug hypersensitivity (Immune system disorders) | 1 | 0 | NA | NA
Appendicitis (Infections and infestations) | 1 | 0 | NA | NA
Bacterial sepsis (Infections and infestations) | 0 | 1 | NA | NA
COVID-19 (Infections and infestations) | 3 | 2 | NA | NA
Cellulitis (Infections and infestations) | 2 | 0 | NA | NA
Dengue fever (Infections and infestations) | 1 | 0 | NA | NA
Diverticulitis (Infections and infestations) | 2 | 0 | NA | NA
Erysipelas (Infections and infestations) | 0 | 2 | NA | NA
Gastroenteritis (Infections and infestations) | 1 | 0 | NA | NA
Infected bite (Infections and infestations) | 1 | 0 | NA | NA
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | NA | NA
Pneumonia (Infections and infestations) | 3 | 1 | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | NA | NA
Urinary tract infection (Infections and infestations) | 2 | 1 | NA | NA
Urosepsis (Infections and infestations) | 0 | 2 | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Fall (Injury, poisoning and procedural complications) | 2 | 1 | NA | NA
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | NA | NA
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Blood ethanol increased (Investigations) | 1 | 0 | NA | NA
Heart rate irregular (Investigations) | 1 | 0 | NA | NA
Hepatic enzyme increased (Investigations) | 0 | 1 | NA | NA
Troponin I increased (Investigations) | 0 | 1 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Lip squamous cell carcinom (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Cerebral infarction (Nervous system disorders) | 0 | 1 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | NA | NA
Ischaemic stroke (Nervous system disorders) | 0 | 3 | NA | NA
Seizure (Nervous system disorders) | 1 | 0 | NA | NA
Syncope (Nervous system disorders) | 4 | 2 | NA | NA
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | NA | NA
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | NA | NA
Haematuria (Renal and urinary disorders) | 1 | 0 | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Period: Placebo (N=178) | Double-blind Period: Patisiran (N=181) | Open Label Extension Period: Placebo (in DB Period) to Patisiran (N=166) | Open Label Extension Period: Patisiran (in DB Period) to Patisiran (N=168)
Cardiac failure (Cardiac disorders) | 68 | 54 | NA | NA
Infusion related reaction (Immune system disorders) | 16 | 22 | NA | NA
Constipation (Gastrointestinal disorders) | 19 | 20 | NA | NA
Atrial fibrillation (Cardiac disorders) | 26 | 16 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 14 | 15 | NA | NA
COVID-19 (Infections and infestations) | 25 | 14 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 14 | NA | NA
Fatigue (General disorders) | 15 | 12 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 12 | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 12 | NA | NA
Gout (Metabolism and nutrition disorders) | 12 | 11 | NA | NA
Fall (Injury, poisoning and procedural complications) | 15 | 10 | NA | NA
Nasopharyngitis (Infections and infestations) | 12 | 10 | NA | NA
Insomnia (Psychiatric disorders) | 11 | 10 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 10 | NA | NA
Dizziness (Nervous system disorders) | 15 | 9 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | NA | NA
Syncope (Nervous system disorders) | 13 | 8 | NA | NA
Nausea (Gastrointestinal disorders) | 9 | 8 | NA | NA
Headache (Nervous system disorders) | 11 | 6 | NA | NA
Orthostatic hypotension (Vascular disorders) | 9 | 3 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is intended that after completion of the study, the data are to be submitted for publication in a scientific journal and/or for reporting at a scientific meeting. A copy of any proposed publication (eg, manuscript, abstracts, oral/slide presentations, book chapters) based on this study, must be provided and confirmed received at the Sponsor at least 30 days before its submission. The Clinical Trial Agreement will detail the procedures for publications.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03997383/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT03997383/SAP_001.pdf